CLINICAL TRIAL: NCT04726475
Title: Impact of Cannabidiol-Rich Hemp Extract Oil on Reconsolidation Disruption of Naturalistic Interoceptive Aversive Memory in Humans
Brief Title: Impact of CBD-Rich Oil on Aversive Memory Reconsolidation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-07-0141
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Anxiety and Fear
MeSH Terms: conditions — Anxiety Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD-WR (Experimental): * 300 mg CBD-rich hemp extract oil administered within the reconsolidation window.
  * The timing of CBD-rich oil administration is based on preclinical studies demonstrating that CBD's disruptive effects on reconsolidation procedurally depend on timing pharmacological administration to be within the memory reconsolidation window (< 6 hrs. post-retrieval).
  * Thus, immediately after the 35% CO2 interoceptive memory reactivation procedure and associated measures (see measures), participants will be asked to take a single 300mg CBD-rich oral dose of a hemp-derived oil formulation.
  Interventions: Behavioral: Interoceptive Aversive Memory Reactivation; Dietary Supplement: Cannabidiol (CBD)-Rich Broad Spectrum Hemp Extract Oil
- PBO-WR (Placebo Comparator): * Placebo administered within the reconsolidation window.
  * Immediately after the 35% CO2 interoceptive memory reactivation procedure and associated measures (see measures), participants will be asked to take a single dose of an MCT coconut oil placebo solution.
  Interventions: Behavioral: Interoceptive Aversive Memory Reactivation; Dietary Supplement: Placebo Oil
- CBD-OR (Active Comparator): * CBD-rich hemp extract oil administered outside of the reconsolidation window.
  * Participants will be asked to take a single 300mg oral dose of CBD-rich oil approximately 24 hrs after the initial 35% CO2 interoceptive memory reactivation challenge.
  * Thus, CBD will be administered well beyond the critical period for memory reconsolidation. The inclusion of this third arm provides a more robust test of the specific reconsolidation theory-based study hypotheses and aids in controlling for any nonspecific possible anxiolytic effects of CBD.
  Interventions: Behavioral: Interoceptive Aversive Memory Reactivation; Dietary Supplement: Cannabidiol (CBD)-Rich Broad Spectrum Hemp Extract Oil

INTERVENTIONS:
Behavioral: Interoceptive Aversive Memory Reactivation — In order to reactivate interoceptive aversive memory, participants will be asked to breathe a medical grade 35% CO2/65% O2 gas mixture which produces somatic perturbations. The 35% CO2 challenge is a widely used and safe symptom induction technique that has been utilized in our laboratory in several experiments. Participants will be informed that breathing the gas is safe, but that it will likely cause changes in their physical sensations. Participants will specifically be asked to breathe the gas mixture normally with their mouth open through an oxygen mask for 10 seconds.
Dietary Supplement: Cannabidiol (CBD)-Rich Broad Spectrum Hemp Extract Oil — 300mg CBD-rich hemp-derived formulation in MCT coconut oil.
  Arms: CBD-OR; CBD-WR
Dietary Supplement: Placebo Oil — 3ml oral dose of MCT coconut oil.
  Arms: PBO-WR

SUMMARY:
The purpose of this study is to test whether cannabidiol (CBD) rich hemp extract oil can interfere with the reconsolidation (storage) of pathological fear memory in humans.

DETAILED DESCRIPTION:
Preclinical experiments demonstrate that isolated cannabidiol (CBD), the non-psychotomimetic constituent of the Cannabis sativa plant, disrupts reconsolidation of aversive memories conditioned in the laboratory when administered within the memory reconsolidation window (< 6 hrs. post-retrieval) by indirectly activating cannabinoid type-1 (CB1) receptors in the dorsal anterior cingulate cortex (dACC). Furthermore, background material (e.g., terpenoids) naturally present in the cannabis plant may also disrupt aversive memory reconsolidation both alone and in concert with CBD. Based on these preclinical findings, we aim to test whether administration of 300mg CBD-rich hemp extract oil following fear reactivation of an aversive interoceptive threat memory can disrupt reconsolidation of naturalistic aversive memories in humans. More specifically, naturalistic interoceptive aversive memories, a form of transdiagnostic fear memory that contributes to the pathogenesis of fear-related disorders such as panic disorder, posttraumatic stress disorder (PTSD), and illness anxiety disorder.

For this proof-of-concept double-blind trial, volunteers (n=96) reporting elevated fears of somatic sensations will be stratified on biological sex and baseline levels of interoceptive fear and randomized to one of three intervention arms: (a). CBD-rich oil administered within the reconsolidation window, (b). Placebo oil administered within the reconsolidation window, or (c). CBD-rich oil administered outside of the reconsolidation window. Change in emotional reactivity to a 35% CO2 challenge from baseline to two-week follow-up will serve as our primary outcome.

Study findings may contribute towards the development of a novel ultra-brief transdiagnostic intervention guided by reconsolidation theory for individuals prone to fear-related psychiatric disorders.

ELIGIBILITY:
Inclusion criteria include:

1. Ages 18-65
2. Fluent in English
3. Willingness to refrain from all non-study cannabis use during the study period.

Exclusion criteria include:

1. Insufficient phobicity (<50 on CO2 challenge);
2. Presence of significant suicidality;
3. History of psychosis;
4. Currently receiving exposure-based treatment;
5. Current substance use disorder;
6. Unstable psychiatric medication for a psychological condition;
7. Medical conditions contraindicating CO2 inhalation (e.g., cardiac arrhythmia, cardiac failure, asthma, lung fibrosis, high blood pressure, epilepsy, or stroke);
8. Any medical problems (e.g., liver or renal abnormalities) or medication use that would preclude ingesting CBD oil, including but not limited to currently taking blood thinners (e.g., Warfarin and some anti-epileptic medications);
9. History of an adverse reaction to CBD oil or other CBD products,
10. Coconut allergy (coconut oil is the carrier oil for CBD-rich extract)

(l) Regular cannabis use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
CO2 Emotional Reactivity | Two-week follow-up
  Self-reported peak-distress (range: 0-100), defined as the highest level of distress experienced at any point during the 35% CO2 challenge completed at the two-week follow-up assessment, adjusting for baseline rating (immediately after the 35% CO2 challenge, but before receiving either immediate CBD/placebo or delayed CBD).

SECONDARY OUTCOMES:
CO2 Emotional Distress Recovery Trajectory | Two-week follow-up
  Participants will be asked to rate their current distress level (range: 0-100) every minute for five consecutive minutes after the CO2 inhalation (recovery phase). Change in CO2 emotional distress recovery trajectory from baseline to the two-week follow will serve as a secondary continuous index of emotional reactivity to somatic cues.
Short Scale Anxiety Sensitivity Index (SASSI) | Two-week
  The 5-item SSASI is a self-report instrument designed to measure the transdiagnostic construct of anxiety sensitivity, defined as a fear of anxiety and arousal-related sensations. Change on the SSASI from baseline to the two-week follow-up will serve as a secondary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Telch, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stern CAJ, de Carvalho CR, Bertoglio LJ, Takahashi RN. Effects of Cannabinoid Drugs on Aversive or Rewarding Drug-Associated Memory Extinction and Reconsolidation. Neuroscience. 2018 Feb 1;370:62-80. doi: 10.1016/j.neuroscience.2017.07.018. Epub 2017 Jul 17. PMID 28729064
- [Background] Murkar A, Kent P, Cayer C, James J, Durst T, Merali Z. Cannabidiol and the Remainder of the Plant Extract Modulate the Effects of Delta9-Tetrahydrocannabinol on Fear Memory Reconsolidation. Front Behav Neurosci. 2019 Aug 1;13:174. doi: 10.3389/fnbeh.2019.00174. eCollection 2019. PMID 31417379
- [Background] Telch MJ, Rosenfield D, Lee HJ, Pai A. Emotional reactivity to a single inhalation of 35% carbon dioxide and its association with later symptoms of posttraumatic stress disorder and anxiety in soldiers deployed to Iraq. Arch Gen Psychiatry. 2012 Nov;69(11):1161-8. doi: 10.1001/archgenpsychiatry.2012.8. PMID 23117637
- [Derived] Zaizar ED, Papini S, O'Connor P, Telch MJ. Impact of cannabidiol-rich hemp extract oil on reconsolidation disruption of naturalistic interoceptive aversive memory in humans: Protocol for a randomized clinical trial. Contemp Clin Trials. 2022 Aug;119:106847. doi: 10.1016/j.cct.2022.106847. Epub 2022 Jul 8. PMID 35811050
- See also: Eligibility survey link — http://telchpsy.co1.qualtrics.com/jfe/form/SV_b9PjqSIzDtzXdNc